CLINICAL TRIAL: NCT00446992
Title: Metabolic Effects of Olanzapine in Patients With Newly Diagnosed Psychosis
Brief Title: Diabetes in Neuropsychiatric Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brian Kirkpatrick, Professor, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK69265; HAC File#: 05-12-141
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizoaffective; psychosis; olanzapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Trial Group (Experimental): The patients were newly diagnosed with psychosis and were recruited at their first clinical contact for psychosis.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — 16-week open trial of olanzapine. The patients were started on a dose of 15 mg/d by mouth, which could be adjusted to as low as 10 mg/d or as high as 40 mg/d, based on clinical response. The trial began while they were hospitalized and continued after discharge.
  Other Names: Zyprexa, Zydis, Relprevv

SUMMARY:
The purpose of this study was to describe metabolic changes in the first 16 weeks of anti-psychotic treatment in previously drug-naïve patients with psychosis.

We hypothesize that in drug-naive patients, greater insulin resistance prior to treatment predicts a disproportionately greater increase in insulin resistance with olanzapine treatment.

DETAILED DESCRIPTION:
Antipsychotic medications are associated with an increased risk of diabetes. We focused on a description of early metabolic adverse effects and clinical and biochemical features that might predict these adverse effects.

ELIGIBILITY:
* Age 18-64
* Maximum cumulative (lifetime) antipsychotic exposure of one week, and no antipsychotic use in the previous 30 days before enrolling in the study
* No history of diabetes or other serious medical or neurological condition associated with glucose intolerance or insulin resistance (eg, Cushing disease),
* Not taking a medication associated with insulin resistance (eg, hydrochlorothiazide, furosemide, ethacrynic acid, metolazone, chlorthalidone), beta blockers, glucocorticoids, phenytoin, nicotinic acid, cyclosporine, pentamidine, or narcotics)
* No history of cocaine use in the previous 30 days, and
* No laboratory evidence of diabetes at baseline (fasting glucose <126 mg/dL or 2-hour glucose <200 mg/dL on a glucose tolerance test)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kirkpatrick, M.D., Principal Investigator — Vice Chair of Psychiatry MCG
Locations (1):
- Unitat Hospitalitzacio - Servei de Psiquiatria G096, Hospital Clinic C/Villarroel, 170, Barcelona, Spain

REFERENCES:
- [Background] Fernandez-Egea E, Miller B, Garcia-Rizo C, Bernardo M, Kirkpatrick B. Metabolic effects of olanzapine in patients with newly diagnosed psychosis. J Clin Psychopharmacol. 2011 Apr;31(2):154-9. doi: 10.1097/JCP.0b013e31820fcea3. PMID 21346617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospital Clinic of Barcelona
Groups:
- Antipsychotic-Naive Patients: The patients were newly diagnosed with psychosis and were recruited at their first clinical contact for psychosis.
  Olanzapine: 16-week open trial of olanzapine. The patients were started on a dose of 15 mg/d by mouth, which could be adjusted to as low as 10 mg/d or as high as 40 mg/d, based on clinical response. The trial began while they were hospitalized and continued after discharge.
Period: Overall Study
Arm/Group | Antipsychotic-Naive Patients
Started | 30 (Beginning of Intervention)
Completed | 14 (Intervention Completion)
Not Completed | 16
Not completed — Adverse Event | 11
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White | 27
  Other | 3
Region of Enrollment [Number; unit: participants]
  Spain | 30
Socioeconomic Status (SES) [Mean (Standard Deviation); unit: units on a scale] — Hollingshead Redlich Scale. Scale: five social classes 1 though 5 (5 being the poorest).
  units on a scale | 4.9 (1.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (3.0)
Number of Cigarettes Per Day [Mean (Standard Deviation); unit: cigarettes per day] | 8.1 (9.7)
Duration of Untreated Psychosis [Mean (Standard Deviation); unit: Months] | 1.5 (1.4)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 82 (8)
Oral Glucose Tolerance Test (OGGT) [Mean (Standard Deviation); unit: mg/dL] — 2-hour, 75-g OGGT, which began between 8 and 9 am after an overnight fast
  mg/dL | 110 (35)
Fasting Insulin [Mean (Standard Deviation); unit: mg/dL] | 9.7 (4.4)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage] | 4.4 (0.3)
Interleukin 6 (IL-6) [Mean (Standard Deviation); unit: pg/mL] | 3.5 (7.2)
Positive and Negative Syndromes Scale (PANSS) [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from a minimum of 30 (not impaired) to a maximum of 210 (greatest impairment) for the total score. Positive, Negative and General scales range from 7 (not impaired) to 49 (greatest impairment), 7 (not impaired) to 49 (greatest impairment), and 16 (not impaired) to 112 (greatest impairment), respectively.
  units on a scale
    PANSS Positive | 25 (7)
    PANSS Negative | 23 (9)
    PANSS General | 39 (10)
    PANSS Total | 87 (20)
C-Reactive Protein [Mean (Standard Deviation); unit: mg/dL] | .21 (.34)
Adiponectin [Mean (Standard Deviation); unit: mg/dL] | 12.3 (5.9)
Leptin [Mean (Standard Deviation); unit: mg/dL] | 7.3 (10.4)
Cortisol [Mean (Standard Deviation); unit: mg/dL] | 18.3 (5.6)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 163 (30)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 80 (26)
LDL [Mean (Standard Deviation); unit: mg/dL] | 97 (27)
HDL [Mean (Standard Deviation); unit: mg/dL] | 50 (14)
Parental History of Type II Diabetes Mellitus [Number; unit: participants]
  Yes | 7
  No | 23

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
kg/m^2
  Baseline | 22.1 (3.0)
  Week 4 | 23.5 (3.2)
  Week 8 | 24.2 (3.0)
  Week 12 | 24.3 (3.0)
  Week 16 | 24.6 (2.7)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p < 0.001, Univariate linear regression

2. Primary Outcome: Fasting Glucose
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
mg/dL
  Baseline | 82.1 (7.7)
  Week 4 | 83.2 (6.8)
  Week 8 | 86.0 (11.0)
  Week 12 | 85.3 (11.1)
  Week 16 | 89.1 (9.9)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = .043, Univariate linear regression

3. Primary Outcome: Fasting Insulin
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
mg/dL
  Baseline | 9.7 (4.4)
  Week 4 | 12.1 (7.6)
  Week 8 | 10.5 (3.2)
  Week 12 | 11.1 (3.0)
  Week 16 | 10.7 (3.3)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = 0.690, Univariate linear regression

4. Primary Outcome: Hemoglobin A1c
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
percentage
  Baseline | 4.4 (.3)
  Week 4 | 4.4 (.2)
  Week 8 | 4.3 (.3)
  Week 12 | 4.4 (.2)
  Week 16 | 4.3 (.2)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = 0.691, Intervariate

5. Primary Outcome: IL-6
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
pg/mL
  Baseline | 3.5 (7.2)
  Week 4 | 3.9 (10.7)
  Week 8 | 6.4 (17.7)
  Week 12 | 3.8 (5.8)
  Week 16 | 2.3 (4.8)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = 0.877, Univariate linear regression

6. Primary Outcome: Triglycerides
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
mg/dL
  Baseline | 80.1 (26.2)
  Week 4 | 98.73 (40.0)
  Week 8 | 107.2 (55.9)
  Week 12 | 115.4 (54.8)
  Week 16 | 113.47 (53.6)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = 0.003, Univariate linear regression

7. Primary Outcome: Cholesterol Total
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
mg/dL
  Baseline | 163.2 (30.1)
  Week 4 | 184.9 (33.3)
  Week 8 | 186.5 (31.4)
  Week 12 | 188.1 (32.9)
  Week 16 | 188.1 (32.9)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = .005, Univariate linear regression

8. Primary Outcome: HDL
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
mg/dL
  Baseline | 49.8 (14.4)
  Week 4 | 50.1 (14.2)
  Week 8 | 49.7 (13.1)
  Week 12 | 49.7 (13.8)
  Week 16 | 48.4 (13.5)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = 0.696, Univariate linear regression

9. Primary Outcome: LDL
Time Frame: Baseline and 4 week intervals
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Trial Group
Number analyzed (Participants) | 30
mg/dL
  Baseline | 96.6 (27.0)
  Week 4 | 115.07 (29.0)
  Week 8 | 116.0 (29.0)
  Week 12 | 116.0 (30.0)
  Week 16 | 117.7 (29.0)
Statistical Analysis 1: Comparison: Open Trial Group; Baseline compared to Week 16; Test type: Superiority or Other; p = 0.013, Univariate linear regression

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Open Follow Up Group: The patients were newly diagnosed with psychosis and this is their first exposure to an antipsychotic.
  Olanzapine: 16-week open trial of olanzapine. The patients were started on a dose of 15 mg/d by mouth, which could be adjusted to as low as 10 mg/d or as high as 40 mg/d, based on clinical response. The trial began while they were hospitalized and continued after discharge.
Arm/Group | Open Follow Up Group
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 11/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Follow Up Group (N=30)
Increased BMI (Metabolism and nutrition disorders) | 9 — Withdrawn because of Exclusion Criteria
Elevated LDL (Vascular disorders) | 2 — Withdrawn because of Exclusion Criteria

LIMITATIONS AND CAVEATS:
The most important limitations in our study were sample size and duration. With a larger sample, some of these measures may have a significant change within this time frame.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No